CLINICAL TRIAL: NCT03364192
Title: Peer-Delivered Whole Health Coaching to Improve Recovery in Veterans With PTSD
Brief Title: Peer-Delivered Whole Health Coaching for Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: D2476-M
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: PTSD
Keywords: Whole Health Coaching; Integrative Health Coaching; Peer Support Specialist; Personalized Health Plan
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: All participants will receive peer-delivered Whole Health Coaching but the start date will be randomized between 4 and 13 weeks from initiation of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Peer-delivered Whole Health Coaching (Experimental): Whole Health Coaching is a Veterans Health Administration variation of integrative health coaching. For this study it will be administered by a peer support specialist.
  Interventions: Behavioral: Whole Health Coaching

INTERVENTIONS:
Behavioral: Whole Health Coaching — Veterans Health Administration variation of integrative health coaching.

SUMMARY:
The investigators are evaluating a service called peer-delivered Whole Health Coaching to understand how it can help Veterans with PTSD. This project has two main goals: (1) determine how peer-delivered Whole Health Coaching can help Veterans with post-traumatic stress disorder and (2) learning about feasibility of implementing this service in Veterans Health Administration primary care settings. The investigators are also evaluating feasibility of the research methods in this trial to learn how to improve future studies on this topic.

Whole Health Coaching is a service designed to improve health and wellness. It is a variation of integrative health coaching and is being used in Veterans Health Administration medical centers. In Whole Health Coaching, Veterans will work with coaches to develop a personal health mission, develop specific goals and action steps, and then adjust their plan as needed. Coaches provide guidance and support throughout the process. In this project, a peer support specialist working in primary care will be the coach. VA Peer Support Specialists, "peers", are Veterans recovering from a mental health condition trained to help other Veterans improve their health.

All participants will receive peer-delivered Whole Health Coaching. Participants will be randomly assigned a start date for their first session with the Peer Whole Health Coach between 4 and 13 weeks after they start the study. The information provided during this time prior to the first session helps us understand how participants do on their own without the service. The research components include interviews and questionnaires about health and wellness, goals, and experiences with the service. Veterans who participate in the study will complete short questionnaires twice a week for 6 months and have four longer appointments where more questions will be asked. Participants will also be given the opportunity to provide feedback on the service.

DETAILED DESCRIPTION:
The investigators are evaluating a service called peer-delivered Whole Health Coaching to understand how it can help Veterans with PTSD. This project has two main goals: (1) determine how peer-delivered Whole Health Coaching can help Veterans with post-traumatic stress disorder and (2) learning about feasibility of implementing this service in Veterans Health Administration primary care settings. The investigators are also evaluating feasibility of the research methods in this trial to learn how to improve future studies on this topic.

Whole Health Coaching is a service designed to improve health and wellness. It is a variation of integrative health coaching and is being used in Veterans Health Administration medical centers. In Whole Health Coaching, Veterans will work with coaches to develop a personal health mission, develop specific goals and action steps, and then adjust their plan as needed. Coaches provide guidance and support throughout the process. In this project, a peer support specialist working in primary care will be the coach. VA Peer Support Specialists, "peers", are Veterans recovering from a mental health condition trained to help other Veterans improve their health.

All participants will receive peer-delivered Whole Health Coaching. Participants will be randomly assigned a start date for their first session with the Peer Whole Health Coach between 4 and 13 weeks after they start the study. The information provided during this time prior to the first session helps us understand how participants do on their own without the service. The research components include interviews and questionnaires about health and wellness, goals, and experiences with the service. Veterans who participate in the study will complete short questionnaires twice a week for 6 months and have four longer appointments where more questions will be asked. Participants will also be given the opportunity to provide feedback on the service.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* Enrolled in primary care at the Syracuse VA (and affiliated CBOCs) and seen in primary care within the past year
* Probable PTSD defined as screening positive for a Criterion A event and PTSD Checklist for DSM-5 (PCL-5) score 33

Exclusion Criteria:

* Unable to communicate in spoken and written English
* Gross cognitive impairment
* Current symptoms of mania/psychosis
* At risk for suicide
* Engaged in psychotherapy in a non-primary care setting
* Changes to psychotropic medications for PTSD within the last 2 months
* Preference for direct referral to specialty mental healthcare

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Johnson, PhD, Principal Investigator — Syracuse VA Medical Center, Syracuse, NY
Locations (1):
- Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Peer-delivered Whole Health Coaching: Whole Health Coaching is a Veterans Health Administration variation of integrative health coaching. For this study it was administered by a peer specialist.
Period: Overall Study
Arm/Group | Peer-delivered Whole Health Coaching
Started | 28
Completed | 12
Not Completed | 16
Not completed — Ineligible | 10
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline information is only available for eligible participants (n = 18). Baseline data is missing for one participant who withdrew following randomization prior to completion of the baseline measures resulting in a sample size of n = 17.
Arm/Group | Peer-delivered Whole Health Coaching
Number analyzed (Participants) | 17
Age, Continuous [Mean (Full Range); unit: years] | 51.71 [28 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Goal Attainment Scaling (GAS)
Description: Goal Attainment Scaling (GAS) is a systematic method used to evaluate participants' individualized goals and progress towards Whole Health goals. Scores range from 0-10 for each domain of whole health measured with higher scores indicating more positive outcomes. Each participant's GAS score reflects the GAS score from the goal domain(s) that the participant identified as primary during the course of the intervention. For participants with multiple goals, GAS scores were average across domains.
Time Frame: Participants completed GAS twice weekly throughout the entire 24 week study period and scores were compared over time.
Population: Participants were included in this analysis if they initiated peer-delivered Whole Health Coaching within 2 weeks of their designated start date, if they met the baseline stability criterion (at least four data points on the primary outcome, the final two of which had to fall within the range of the previous two data points, for at least 5 of the 9 domains), and if they completed at least three assessments during the intervention phase.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Peer-delivered Whole Health Coaching: Whole Health Coaching is a Veterans Health Administration variation of integrative health coaching. For this study it was administered by a peer support specialist.
Arm/Group | Peer-delivered Whole Health Coaching
Number analyzed (Participants) | 10
score on a scale
  Baseline Phase | 2.33 (0.90)
  Peer-Delivered Whole Health Coaching Phase | 4.15 (0.75)
  Maintenance/Follow-up Phase | 4.63 (1.09)
Statistical Analysis 1: Comparison: Peer-delivered Whole Health Coaching; Test type: Other — Multilevel modeling adapted for multiple-baseline design comparing participant goal attainment before, during, and after peer-delivered Whole Health Coaching; p < 0.05, Multilevel Modeling

2. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: The PTSD Checklist for DSM-5 (PCL-5) is a measure of participants' PTSD symptoms. The total sum score ranges from 0-80 with lower scores indicating more positive outcomes.
Time Frame: Participants completed the PCL-5 at baseline, pre-treatment, post-treatment, and final follow-up assessments over the course of the 24 week study period.
Population: Only participants included in the primary analysis are analyzed here.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Peer-delivered Whole Health Coaching
Number analyzed (Participants) | 10
score on a scale
  Baseline | 42.4 (4.40)
  Before Peer-Delivered Whole Health Coaching | 53.5 (4.40)
  After Peer-Delivered Whole Health Coaching | 49.22 (4.67)
  Follow-up (24 weeks) | 49.61 (4.67)

3. Secondary Outcome: Inventory of Psychosocial Functioning (IPF)
Description: The Inventory of Psychosocial Functioning (IPF) is a measure of psychosocial functioning across several domains. The total score was used for this project and reflects a composite of multiple subscales (romantic relationships, family, work, friendships and socializing, parenting, education, and self care). Scores range from 0-100 with lower scores indicating more positive outcomes.
Time Frame: Participants completed the IPF at baseline, pre-treatment, post-treatment, and final follow-up assessments over the course of the 24 week study period.
Population: Only participants meeting criteria for inclusion in the primary analysis are included here.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Peer-delivered Whole Health Coaching
Number analyzed (Participants) | 10
score on a scale
  Baseline | 38.74 (4.54)
  Before Peer-Delivered Whole Health Coaching | 30.49 (4.54)
  After Peer-Delivered Whole Health Coaching | 28.24 (4.77)
  Follow-Up (24 weeks) | 28.59 (4.77)

4. Secondary Outcome: Client Satisfaction Questionnaire
Description: Measure of participants' satisfaction with the peer-delivered Whole Health Coaching service. CSQ-8 scores range from 8-32 with higher values indicating more positive outcomes.
Time Frame: 8 weeks following intervention onset
Population: The CSQ-8 was analyzed for all participants with non-missing data at this timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Peer-delivered Whole Health Coaching
Number analyzed (Participants) | 11
score on a scale | 27.18 (4.07)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Peer-delivered Whole Health Coaching
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peer-delivered Whole Health Coaching (N=18)
Non-Serious Adverse Event-Unrelated to Study Participation (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT03364192/Prot_SAP_000.pdf